CLINICAL TRIAL: NCT01552109
Title: STable Angina obseRvational Registry
Acronym: STAR
Status: Completed | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 10037399DOC
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Stable Angina
Keywords: symptomatic stable angina; subjects with symptomatic stable angina visiting non-interventional consulting physicians for treatment and meets the inclusion/exclusion criteria
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the clinical profile and current status of the diagnosis and management of stable angina in India by non-interventional consulting physicians (CP) through a large multicenter observational registry.

DETAILED DESCRIPTION:
An observational registry on diagnosis and management of stable angina in India Purpose To describe the clinical profile and current status of the diagnosis and management of stable angina in India by non-interventional consulting physicians (CP) through a large multicenter observational registry.

Design A prospective, multi-center, observational registry. Subject Population Adult, male or female subjects with symptomatic stable angina visiting non-interventional consulting physicians for treatment and who meet the study inclusion/exclusion criteria.

Enrollment:

The study is expected to enroll 1000 to 1500 subjects by 150 - 250 non-interventional consulting physicians. The enrollment period will be around 4 months.

Inclusion criteria

Subject must meet all of the following criteria to be eligible for inclusion in the trial:

1. Subject has been provisionally diagnosed with stable angina by the CP (consulting physician) during the current visit or within 3 months preceding the current visit
2. Subject agrees to sign a data release form

Exclusion criteria

Subjects will be excluded from the trial if any of the following criteria are met:

1. Subject has a history of Acute Coronary Syndrome
2. Subject has a history of prior revascularization
3. Subject has a history of previous MI
4. Subject has new onset angina with symptoms less than one month

Objectives:

1. Describe the demographic and medical profile of subjects diagnosed with stable angina by non-interventional consulting physicians in India
2. Describe the diagnostic pathway prescribed by non-interventional consulting physicians and adopted by stable angina subjects in India
3. Describe the management of stable angina by non-interventional consulting physicians and undertaken by subjects in India

ELIGIBILITY:
Inclusion criteria

Subject must meet all of the following criteria to be eligible for inclusion in the trial:

1. Subject has been provisionally diagnosed with stable angina by the CP (consulting physician) during the current visit or within 3 months preceding the current visit
2. Subject agrees to sign a data release form

Exclusion criteria

Subjects will be excluded from the trial if any of the following criteria are met:

1. Subject has a history of Acute Coronary Syndrome
2. Subject has a history of prior revascularization
3. Subject has a history of previous MI
4. Subject has new onset angina with symptoms less than one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, male or female subjects with symptomatic stable angina visiting non-interventional consulting physicians for treatment and who meet the study inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2079 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- East Delhi Clinic, New Delhi, New Delhi, India